CLINICAL TRIAL: NCT04763772
Title: Clinical Effectiveness of Body Fat Distribution Imaging in Real-World Practice: The BODY-REAL Study
Acronym: BODY-REAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Ian J. Neeland, MD, Director, UH Center for Cardiovascular Prevention, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20201918
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity; PreDiabetes; Type 2 Diabetes; Cardiovascular Risk Factor
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Detailed Report (Experimental): A detailed body composition profile report that consists of the following elements: basic demographic data, percent body fat, weight to muscle ratio, visceral fat and abdominal subcutaneous fat volume, visceral fat ratio (the fraction of visceral divided by total abdominal fat), muscle fat infiltration and liver fat (%), and thigh muscle volumes (also separated into right and left, anterior and posterior compartments). Each parameter is presented on a visual scale in the context of the individual value, general population defined by reference data (from United Kingdom (UK) Biobank population), a metabolic disease-free population (also from UK Biobank), low/high and very low/very high, corresponding to 15th and 5th percentiles, respectively. There are also descriptions of each biomarker and how they are derived to provide context for the recipient.
  Interventions: Diagnostic Test: Body Fat Distribution Imaging Report
- Basic Weight Information (Placebo Comparator): A simple informational report consisting of weight, BMI, and a visual representation of their BMI. This report also categorizes their BMI into underweight, normal weight, overweight, or obese categories according to the World Health Organization categorization schema.
  Interventions: Diagnostic Test: Basic Weight Information
- Patient Provided (Experimental): Report provided directly to the patient.
  Interventions: Behavioral: Patient Provided
- Physician Provided (Placebo Comparator): Report provided directly to the provider to translate/counsel the patient.
  Interventions: Behavioral: Physician Provided

INTERVENTIONS:
Diagnostic Test: Body Fat Distribution Imaging Report — Those randomized to body fat distribution imaging will be scanned on a 1.5 Tesla Siemens Aera MRI scanner (Siemens, Erlangen, Germany), located in the Center for Advanced Heart and Vascular Care using a 6-minute dual-echo Dixon Vibe protocol providing a water and fat separated volumetric data set covering neck to knees, and a multiecho Dixon acquisition for proton density fat fraction assessment in the liver. Images of the liver will be acquired using a 16-channel SENSE extra large Torso coil and images from the rest of the body will be acquired using the body coil. Volumetric imaging datasets of the body derived by MRI will be generated and adipose tissue/fat depots will be quantified: abdominal subcutaneous compartment (ASAT), visceral compartment (VAT), and hips and buttocks (lower body fat); proton density fat fraction of the liver (i.e. hepatic steatosis) as well as the quality of lean (skeletal muscle) including muscle volume and degree of fat infiltration.
  Arms: Detailed Report
Diagnostic Test: Basic Weight Information — Body weight and body mass index
  Arms: Basic Weight Information
Behavioral: Patient Provided — Body weight/fat distribution information will be provided directly to the patient
  Arms: Patient Provided
Behavioral: Physician Provided — Body weight/fat distribution information will be provided directly to the physician
  Arms: Physician Provided

SUMMARY:
The overall goal is to determine the real-world feasibility and utility of body fat imaging using rapid MRI to enhance risk perception, induce behavioral change, and improve clinical outcomes in overweight and obese individuals. Here, the investigators will perform a pragmatic clinical effectiveness pilot trial using a 2x2 factorial design to test the hypothesis that provision of a detailed individualized visual report of body fat distribution directly to patients will translate into changes in patient risk perception, behavior, and improved clinical outcomes.

DETAILED DESCRIPTION:
Specific Aim 1: To compare the clinical effectiveness of communicating the body weight and BMI using a visual aid alone versus a detailed body fat distribution report including individualized images and values relative to normative data using a visual scale in a population of overweight and obese adults with prediabetes or type 2 diabetes and at least one additional cardiovascular disease risk factor. Hypothesis 1: Provision of a detailed body fat distribution report contextualized with information describing the relevance of each body fat parameter will be superior to provision of body weight/BMI information alone on risk perception, behavioral change (enhanced physical activity, dietary choices, and preventive provider practices and medication adherence), and clinical outcomes (reduction in weight and waist circumference, blood pressure, triglycerides, and glycosylated hemoglobin).

Specific Aim 2: To compare the clinical effectiveness of communicating body fat information to the medical provider (with the intent that the provider interprets the data and translates it to the patient) versus communicating the body fat information directly to the patient. Hypothesis 2: Provision of body fat information directly to the patient will be superior to provision of the information to the provider on risk perception, behavioral change, and clinical outcomes (as assessed in Aim 1).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 35 years
2. Able to provide informed consent
3. Overweight or Obese (BMI ≥25 kg/m2)
4. Prediabetes or Type 2 Diabetes:

   * Fasting glucose >100 mg/dl, or
   * Hb A1c >5.7%, or
   * Medical (i.e. pharmacologic) treatment for type 2 diabetes
5. At least 1 additional cardiovascular risk factor (defined by Adult Treatment Panel III criteria2) including:

   * Hypertension (BP>130/80 or on medical therapy for hypertension)
   * Low HDL-cholesterol (<40 mg/dL in men and <50 mg/dL in women)
   * High triglycerides (>150 mg/dL or on treatment for hypertriglyceridemia)
   * Obstructive sleep apnea (clinical diagnosis)
   * Coronary artery disease (clinical diagnosis)
   * Congestive heart failure (clinical diagnosis)
   * Atrial fibrillation (clinical diagnosis)

Exclusion Criteria:

1. Receipt of any anti-obesity drug or supplement within 1 month prior to screening for this trial or plan to initiate therapy during the trial.
2. Self-reported or clinically documented history of significant fluctuations (>5% change) in weight within 1 month prior to screening for this trial.
3. Current or history of treatment with medications that may cause significant weight gain, within 1 month prior to screening for this trial, including systemic corticosteroids (except for a short course of treatment, i.e., 7- 10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g., imipramine, amitryptiline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium).
4. Surgery scheduled for the trial duration period, except for minor surgical procedures, at the discretion of the Investigator.
5. Language barrier, mental incapacity, unwillingness or inability to understand.
6. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods. These include abstinence and the following methods: diaphragm with spermicide, condom with spermicide (by male partner), intrauterine device, sponge, spermicide, Norplant®, Depo-Provera® or oral contraceptives.
7. Unable to complete/tolerate magnetic resonance imaging (MRI) due to severe claustrophobia or metallic implants.
8. ≥2 no-shows to recruitment clinic within the 6 months prior to screening.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this proposed research application will be available to other researchers both internally at University Hospitals/Case Western Reserve University and externally at other institutions. All data will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects. For external researchers, a similar procedure will be required in addition to signing a Data Use and Distribution Agreement per standard University policies and procedures. Data sharing will be in accordance with Institutional policies, local Institutional Review Board (IRB) rules, as well as local, state and Federal laws and regulations, including the HIPAA Privacy Rule.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately after study publication for 2 years

REFERENCES:
- [Derived] Chhabria SM, Perez JA, Neeland IJ. Impact of an MRI Body Fat Imaging Report on Obesity-Related Cardiometabolic Risk: Findings From the BODY-REAL Study, A Randomized Trial. Obes Sci Pract. 2025 Nov 12;11(6):e70099. doi: 10.1002/osp4.70099. eCollection 2025 Dec. PMID 41245699

RESULTS

PARTICIPANT FLOW:
Groups:
- Detailed Report + Patient Provided: A detailed read-out of body fat and muscle quantitation and distribution including visceral fat, abdominal subcutaneous fat, and thigh muscle volumes in liters, and thigh muscle fat infiltration (%) and liver fat (%), all presented on a visual scale compared with reference data from a normative, metabolic disease-free population (derived from the UK Biobank).
  Report provided to the patient.
- Basic Weight Information + Patient: A simple informational report consisting of weight, BMI, and a visual representation of their BMI. This report also categorizes their BMI into underweight, normal weight, overweight, or obese categories according to the World Health Organization categorization schema.
  Basic Weight Information: Body weight and body mass index
  Report provided to the patient.
- Detailed Report + Doctor Provided: A detailed read-out of body fat and muscle quantitation and distribution including visceral fat, abdominal subcutaneous fat, and thigh muscle volumes in liters, and thigh muscle fat infiltration (%) and liver fat (%), all presented on a visual scale compared with reference data from a normative, metabolic disease-free population (derived from the UK Biobank).
  Report provided to medical professional.
- Basic Weight Information + Doctor Provided: A simple informational report consisting of weight, BMI, and a visual representation of their BMI. This report also categorizes their BMI into underweight, normal weight, overweight, or obese categories according to the World Health Organization categorization schema.
  Basic Weight Information: Body weight and body mass index
  Report provided to medical professional.
Period: Overall Study
Arm/Group | Detailed Report + Patient Provided | Basic Weight Information + Patient | Detailed Report + Doctor Provided | Basic Weight Information + Doctor Provided
Started | 6 | 8 | 8 | 7
Completed | 6 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detailed Report + Patient Provided | Basic Weight Information + Patient | Detailed Report + Doctor Provided | Basic Weight Information + Doctor Provided | Total
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.0) | 60.5 (13.9) | 66.0 (9.9) | 64.3 (8.7) | 63.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 1 | 9
  Male | 5 | 5 | 4 | 6 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 8 | 7 | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.2 (3.1) | 35.1 (6.3) | 31.5 (4.9) | 35.5 (8.3) | 33.6 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI
Description: Change in body mass index between groups
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | Detailed Report + Patient Provided | Basic Weight Information + Patient | Detailed Report + Doctor Provided | Basic Weight Information + Doctor Provided
Number analyzed (Participants) | 6 | 8 | 8 | 7
kg/m2 | 0.43 [-6.3 to 7.2] | 0 [0 to 0] | 4.4 [-2.0 to 11] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Detailed Report + Patient Provided vs Basic Weight Information + Patient vs Detailed Report + Doctor Provided vs Basic Weight Information + Doctor Provided; Test type: Superiority; p = 0.2, Regression, Linear; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-14 to 4.8]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Detailed Report + Patient Provided | Basic Weight Information + Patient | Detailed Report + Doctor Provided | Basic Weight Information + Doctor Provided
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04763772/Prot_SAP_001.pdf